CLINICAL TRIAL: NCT05466474
Title: A Single-center, Open-arm, Single-arm Phase II Trial of the PD-1 Antibody Tirelizumab Plus Dacarbazine as First-line Treatment for Advanced Melanoma
Brief Title: PD-1 Antibody Tislelizumab Combined With Dacarbazine in the Treatment of Advanced Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, Associate chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZUSC-13
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-09

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — tislelizumab; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with dacarbazine (Experimental): Tislelizumab combined with dacarbazine in the treatment of advanced melanoma.
  Interventions: Biological: Tislelizumab Injection

INTERVENTIONS:
Biological: Tislelizumab Injection — Efficacy of tislelizumab or tislelizumab combined with dacarbazine in the treatment of advanced malignant melanoma.
  Other Names: Dacarbazine

SUMMARY:
A total of 40 subjects who had not received systemic treatment or chemotherapy in the past and were allowed to receive adjuvant or neoadjuvant treatment for advanced melanoma received tirelizumab combined with dacarbazine for 4-6 cycles to evaluate the efficacy, safety and prognosis of tirelizumab combined with dacarbazine in the treatment of advanced melanoma.

DETAILED DESCRIPTION:
In henan province tumor hospital into the group of 40 cases always will not accept any systemic therapy or chemotherapy, allowed to always have a recurrence of adjuvant or neoadjuvant therapy sensitive sensitive relapse (referring to more than six months after the last chemotherapy recurrence) of unresectable melanoma metastatic/operation subjects, accept for LeiLiZhu a joint resistance of kappa oxazine treatment 4-6 cycles, To evaluate the efficacy, safety and prognosis of tislelizumab combined with dacarbazine in the treatment of advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-72 years (inclusive);
2. patients with unresectable stage III or IV melanoma diagnosed histologically or cytologically;
3. According to the efficacy evaluation criteria for solid tumors (RECIST V1.1), there are lesions that can be used as target lesions for evaluation;
4. Prior adjuvant or neoadjuvant therapy must have been completed for at least 4 weeks prior to study drug administration, and all associated toxic effects (except hair loss) have been recovered (to ≤ class 1 or baseline) prior to study drug administration;
5. ECOG score was 0-1;
6. The expected survival time is more than 3 months;
7. No major surgery (except for baseline tumor biopsy) or severe trauma occurred at least 14 days prior to the first administration of study therapy;
8. Adequate organ and bone marrow function, as defined below:

   Blood routine (no blood transfusion, no G-CSF, no drug correction within 14 days prior to screening) Neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 109 /L); Platelet count (PLT) ≥ 100,000/mm3 (100 × 109 /L); Hemoglobin (Hb) ≥ 9 g/dL (90 g/L); Blood biochemical Serum creatinine (Cr) ≤ 1.5× upper limit of normal (ULN) or creatinine clearance Rate (Cockroft-Gault formula) ≥ 60 mL /min; Total bilirubin (TBIL) ≤ 1.5×ULN; Aspartate aminotransferase (AST) or ALT ≤2.5×ULN, Subjects with liver metastasis should be ≤5×ULN; Blood coagulation function International standardized ratio (INR) ≤1.5, prothrombin time (PT) and Activated partial thrombin time (APTT) ≤1.5×ULN; Routine urine urinary protein <2+; If urinary protein ≥2+, 24 hours of urinary protein quantitative significant Protein must be ≤1g; Thyroid function Thyroid stimulating hormone (TSH) ≤ ULN; If abnormal, FT3(T3) should be investigated.

   And FT4(T4), and normal FT3(T3) and FT4(T4) levels could be selected;
9. Female subjects of reproductive age must have performed a serological pregnancy test within 7 days prior to medication, with negative results, and be willing to use a medically approved highly effective contraceptive method (e.g., an intrauterine device, birth control pill, or condom) during the study period and for 3 months after the last medication; For male subjects with a female partner of reproductive age, surgical sterilization or consent was required during and after the study
10. Able to understand and voluntarily sign written informed consent;
11. Subjects must be willing and able to complete study procedures and follow-up examinations.

Exclusion Criteria:

1. Prior treatment with anti-PD-1, anti-PD-L1, and anti-PD-L2;
2. Previous treatment with dacarbazine
3. Received any other study treatment within 4 weeks prior to C1D1;
4. Surgical treatment and/or radiation therapy for melanoma are planned during the study period.
5. Imaging diagnosis showed the presence of central nervous system tumor lesions.
6. prior use of immunosuppressive drugs within 14 days prior to C1D1, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (i.e., no more than 10mg/ day of prednisone or other corticosteroids at pharmacologically equivalent doses).
7. The presence or history of any active autoimmune diseases (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or asthma that was in complete remission during childhood and did not currently require medical intervention could be included), or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
8. Severe infection (e.g., antibiotic, antifungal, or antiviral medication) within 4 weeks prior to C1D1, or unexplained fever >38.5°C during screening/prior to initial administration.
9. Significant clinical bleeding symptoms or clear bleeding tendency occurred within 3 months before C1D1, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occultation blood ++ or above, vasculitis, etc.; Or arteriovenous thrombosis events occurring within 6 months prior to C1D1, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.; Or long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300mg/ day or clopidogrel ≥75mg/ day).
10. Active heart disease, including myocardial infarction, severe/unstable angina, etc., within 6 months before C1D1. Arrhythmias with poorly controlled left ventricular ejection fraction <50% on echocardiography (including QTcF interval >450ms in men and >470ms in women).
11. C1D1 has been diagnosed with any other malignancy within the previous 5 years, except for adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix.
12. known allergy to the study drug or any excipients thereof; Or severe allergic reactions to other monoclonal antibodies.
13. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B surface antigen positive and HBV-DNA ≥500IU/ mL), hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the detection limit of analysis method).
14. In the judgment of the investigator, there are concomitants (such as poorly controlled hypertension, severe diabetes, neurological or neurologic diseases, etc.) or any other conditions that seriously endanger the safety of the subjects, may confuse the results of the study, or may interfere with the completion of the study.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to approximately 24months
  Until the tumor progresses or the patient dies or is lost to follow-up or cannot tolerate it
Progression-free survival | Up to approximately 24months
  From the start of treatment to the onset of disease progression or death of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No